CLINICAL TRIAL: NCT06110377
Title: MALE ANDROGENETIC ALOPECIA - Treatment With Dutasteride Injections: Mesotherapy (Injections With Syringe and Needle) x MMP Technique (Microinjections With Tattoo Machine)
Brief Title: MALE HAIR LOSS - Treatment With Dutasteride Mesotherapy x Dutasteride MMP Technique (Injections With Tattoo Machine)
Acronym: MMP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Dermatologica Arbache ltda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2023-10-22; First posted 2023-10-31 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Androgenic Alopecia
Keywords: Dutasteride; Administration, Cutaneous; Mesotherapy
MeSH Terms: conditions — Alopecia | interventions — Mesotherapy; Injections; Syringes; Needles; Matrix Metalloproteinases

STUDY DESIGN:
Intervention Model Description: This is a randomized study carried out on 60 men. Two techniques for administering dutasteride will be compared, injected by syringes or needles (mesotherapy) or needling using the MMP technique (through tattoo machines)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MESOTHERAPY (INJECTIONS WITH SYRINGE AND NEEDLE) (Active Comparator): After the anesthetic block, dutasteride will be injected using syringes and needles into the area of alopecia.
  Interventions: Procedure: MESOTHERAPY (INJECTIONS WITH SYRINGE AND NEEDLE)
- MMP (INJECTIONS WITH TATTOO MACHINE) (Experimental): After the anesthetic block, dutasteride will be injected through needling performed by a tattoo machine in the area of alopecia.
  Interventions: Procedure: MMP (INJECTIONS WITH A TATTOO MACHINE)

INTERVENTIONS:
Procedure: MESOTHERAPY (INJECTIONS WITH SYRINGE AND NEEDLE) — After the anesthetic block, dutasteride will be injected using syringes and needles into the area of alopecia.
  Arms: MESOTHERAPY (INJECTIONS WITH SYRINGE AND NEEDLE)
Procedure: MMP (INJECTIONS WITH A TATTOO MACHINE) — After the anesthetic block, dutasteride will be injected through needling performed by a tattoo machine in the area of alopecia.
  Arms: MMP (INJECTIONS WITH TATTOO MACHINE)

SUMMARY:
This randomized clinical trial carried out on 60 Brazilian men, aged 18 to 65, with mild or moderate androgenetic alopecia. Two techniques for administering dutasteride will be compared, injected by syringes or needles or by needling through tattoo machines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers male patients.
* Aged 18 to 65 years.
* Patients with male androgenetic alopecia (grades III - V of the Norwood/Hamilton scale)
* Commitment not to initiate any other treatment, topical, systemic or intralesional, that interferes with hair growth during the study period.
* Patient without systemic treatment for AGA (5 reductase inhibitors) for more than 12 months or without topical treatment for more than 6 months before the start of the study.
* Allow the creation of two micro tattoos (maximum size of 1 mm each, resembling a hairy infundibulum) in the area that will be treated, in order to standardize the trichoscopic analysis.
* With the aim of photographic standardization, the patient must agree to have their hair cut in a standardized way in the first and last interventions.
* Patient about to get his partner pregnant.
* Patient must refrain from donating blood during the investigation and up to 6 months after the last intervention,
* Patient must abstain from drinking alcoholic beverages, abstain from using inhaled or injectable drugs, abstain from using illicit drugs within 30 days of entering the study,
* Patients without a psychiatric diagnosis and who behave appropriately during the interview,
* Signs of good hygiene and that have the ability to keep the areas undergoing treatment clean until they heal,
* Patients who understand and speak Portuguese,
* Patients with realistic expectations regarding the final benefits of treatment,
* Needle phobia,
* Independent patient, eliminating the need for tutoring or legal representative,
* Absence of chronic viral diseases, for example HIV, hepatitis B or hepatitis C,
* Absence of other skin diseases, for example lichen planus, psoriasis, Crohn's disease or ulcerative colitis,
* Absence of immunosuppression, for example: lymphoma, transplant therapy, chronic corticosteroid use, Wiskott-Aldrich Syndrome or uncontrolled malignancy,
* Patients/participants with previously known allergies or those detected during the interventions (anesthetics, topical antibiotics or other medications used in the trials),
* Absence of clinically significant cardiovascular disease (e.g. previous myocardial infarction), absence of coagulopathy or use of anticoagulants, absence of neurological disease (e.g. stroke, cerebral ischemia), absence of renal, hepatic or endocrine disease (e.g. example, diabetes).
* Patient/participant with medical conditions not mentioned, which in the investigator's view, prohibit participation in the study.
* Signature of informed consent

Exclusion Criteria:

* Detection during the test of allergy to the medicines used (anesthetics, topical antibiotics or other medicines used in the tests),
* Breach of protocol, inappropriate conduct that compromises participant safety or interferes with the interpretation of study results,
* Any illness or condition, which in the judgment of the investigators, interferes with the participant's ability to complete or terminate the investigation.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — yes
Enrollment: 60 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
HAIR DENSITY | 1 year
  analysis of hair density (number of follicles) per square centimeter using Trichoscale software (fotofinder) and clinical photographs.
HAIR THICKNESS | 1 year
  measurement of the thickness of hair shafts using Trichoscale software (fotofinder)

SECONDARY OUTCOMES:
Sexual effects | 1 year
  Assessment of sexual adverse effects (sexual impotence or decreased libido) through Likert questionnaire: The answer will be dichotomous, did you feel any sexual effects (impotence or decreased libido during your treatment? Yes or no?

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Dermatologica Arbache, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No